CLINICAL TRIAL: NCT00945035
Title: An Open-Label, Randomized, 2-Period, Single-Dose, Balanced, Crossover Study in Healthy Subjects to Establish the Bioequivalence of the 20% and 30% Etoricoxib (MK0663) Formulations
Brief Title: Study of the Bioequivalence of the 20% and 30% Etoricoxib Tablet Formulations (0663-070)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0663-070; MK0663-070; 2009_623
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Etoricoxib

ARMS (2):
- A (Active Comparator): Etoricoxib, 20% tablet
  Interventions: Drug: etoricoxib
- B (Active Comparator): Etoricoxib, 30% tablet
  Interventions: Drug: Comparator: etoricoxib

INTERVENTIONS:
Drug: etoricoxib — Single dose etoricoxib 120 mg 20% final market image tablet in one of two treatment periods.
  Arms: A
Drug: Comparator: etoricoxib — Single dose etoricoxib 120 mg 30% unmilled, roller compaction tablet in one of two treatment periods.
  Arms: B

SUMMARY:
This study will establish the bioequivalence of the 20%, milled, roller compaction final market image (FMI) etoricoxib tablets and 30% unmilled, roller compaction (UMC) etoricoxib tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subject is in good health
* Subject agrees to follow the study guidelines

Exclusion Criteria:

* Subject is a smoker
* Subject has a history of adverse reactions caused by NSAIDs or allergies/intolerance to NSAIDs
* Subject is in a situation or has a condition/disease which may interfere with optimal participation in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2002-11; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Etoricoxib FMI Then Etoricoxib URC: FMI Formulation (20%), Final Market Image/ URC Formulation (30%), Unmilled Roller Compaction
- Etoricoxib URC Then Etoricoxib FMI: URC Formulation (30%), Unmilled Roller Compaction/ FMI Formulation (20%), Final Market Image
Period: Period 1
Arm/Group | Etoricoxib FMI Then Etoricoxib URC | Etoricoxib URC Then Etoricoxib FMI
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Etoricoxib FMI Then Etoricoxib URC | Etoricoxib URC Then Etoricoxib FMI
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants in Study
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: Years] | 36.1 [18 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 19
Height [Mean (Full Range); unit: Centimeters] | 168.3 [149.9 to 193.0]
Weight [Mean (Full Range); unit: Kilograms] | 75.2 [50.5 to 99.1]

OUTCOME MEASURES:

1. Primary Outcome: Plasma Area Under the Curve (AUC(0 to Infinity)) for Etoricoxib
Description: The area under the plasma concentration vs time curve.
Time Frame: Through 120 Hours Postdose
Population: All healthy adult subjects completed the study and were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: µg times hr/mL
Groups:
- Etoricoxib FMI: FMI Formulation (20%), Final Market Image.
- Etoricoxib URC: URC Formulation (30%), Unmilled Roller Compaction
Arm/Group | Etoricoxib FMI | Etoricoxib URC
Number analyzed (Participants) | 36 | 36
µg times hr/mL | 32.65 (16.20) | 33.28 (13.65)
Statistical Analysis 1: Comparison: Etoricoxib FMI vs Etoricoxib URC; Least-Squares Mean Ratio (B/A); A=FMI Formulation (20%), Final Market Image; B=URC Formulation (30%), Unmilled Roller Compaction; Test type: Non-Inferiority or Equivalence — Study Primary Hypothesis: The plasma etoricoxib AUC(0-∞) and Cmax values following a single-dose administration of the 120 mg etoricoxib (30%) URC formulation will be bioequivalent to the plasma AUC(0-∞) and Cmax of 120 mg etoricoxib (20%) in the FMI formulation following single-dose administration (geometric mean ratio [GMR] no less than 0.8 and no greater than 1.25); Least-Squares Mean Ratio = 1.02, 90% CI [0.97 to 1.07]

2. Primary Outcome: Peak Plasma Concentration (Cmax) for Etoricoxib
Time Frame: Through 120 Hours Postdose
Population: All healthy adult subjects completed the study and were included in the statistical analysis.
Measure: Least Squares Mean (Standard Deviation); unit: ng/mL
Arm/Group | Etoricoxib FMI | Etoricoxib URC
Number analyzed (Participants) | 36 | 36
ng/mL | 1964 (701) | 2021 (833)
Statistical Analysis 1: Comparison: Etoricoxib FMI vs Etoricoxib URC; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Least-Squares Mean Ratio = 1.03, 90% CI [0.95 to 1.11]

ADVERSE EVENTS:
Description: Although a subject/patient may have had two or more clinical adverse experiences, the subject/patient is counted only once within a category. The same subject/patient may appear in different categories.
Arm/Group | Etoricoxib FMI | Etoricoxib URC
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36
Other Adverse Events (participants affected / at risk) | 9/36 | 12/36
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etoricoxib FMI (N=36) | Etoricoxib URC (N=36)
Dry Mouth (Gastrointestinal disorders) | 1 | 2
Loose Stools (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 6 | 7
Headache (Nervous system disorders) | 1 | 3
Somnolence (Nervous system disorders) | 3 | 4
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.